CLINICAL TRIAL: NCT01530776
Title: Preventing Postpartum Weight Retention Among Low-Income, Black Women
Brief Title: Healthy4Baby: Preventing Postpartum Weight Retention Among Low-Income, Black Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20227; K23HL106231 (NIH)
Record Dates: First submitted 2012-01-23; First posted 2012-02-10 (Estimated); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Pregnancy; Weight Loss; Behavioral; Obesity
Keywords: Pregnancy; Postpartum; Weight Retention; Behavioral; Electronically-mediated
MeSH Terms: conditions — Weight Loss; Behavior; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy Lifestyle Group (Experimental): Participants randomized to this condition will receive information and strategies to help them eat healthier and be more active during and after pregnancy. They will get this information about eating and activity through handouts, text messages, Facebook updates, and in-person visits and phone calls from a health coach.
  Interventions: Behavioral: Healthy Lifestyle Group
- Usual Care (No Intervention): This condition is meant to represent standard clinical care provided to pregnant and postpartum mothers at Temple University.

INTERVENTIONS:
Behavioral: Healthy Lifestyle Group — Electronically-mediated, behavioral intervention during and after pregnancy encouraging mothers to eat healthy, exercise, and return to their early pregnancy weights by 1 year postpartum
  Arms: Healthy Lifestyle Group

SUMMARY:
The purpose of this study is to assess the feasibility and efficacy of an electronically-mediated, pregnancy and postpartum, behavioral intervention program, compared to usual obstetric care, on changes in weight and cardiometabolic biomarkers among overweight and obese Black women.

DETAILED DESCRIPTION:
Black women are in particular need for obesity prevention and treatment. Targeting the childbearing period has the potential to slow the accumulation of weight gain among this high risk group. Previous interventions to prevent postpartum weight retention among Blacks are sparse and limited by poor intervention adherence, high attrition, and failure to include pregnancy in the study design. The proposed research aims to overcome these shortcomings by developing an intervention that 1) focuses solely on Black women, 2) incorporates Black mothers' information needs, values, and social context, 3) uses technology to facilitate participant engagement, and 4) includes both the pregnancy and postpartum periods.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant African-American women at least 18 years of age
2. BMI at recruitment between 25.0-44.9 kg/m2
3. Singleton pregnancy
4. Gestational age of ≤ 20 weeks as determined by last menstrual period
5. Plan to carry the pregnancy to term and keep the baby
6. Own a cell phone with a text messaging plan
7. Member of Facebook social networking site
8. Able to participate in physical activity
9. Participants must be willing to comply with all study-related procedures

Exclusion Criteria:

1. BMI ≤ 24.9 or ≥ 45.0
2. Uncontrolled hypertension (systolic blood pressure > 160 or diastolic blood pressure > 95 mmHg). Participants with controlled hypertension on medication for at least three months are allowable.
3. Known atherosclerotic cardiovascular disease
4. Known congestive heart failure
5. Known diabetes mellitus (type 1 or type 2)
6. Uncontrolled thyroid disease. Participants with controlled thyroid disease on medication for at least three months are allowable.
7. Known cancer
8. Any major active rheumatologic, pulmonary, hepatic, dermatologic disease or inflammatory condition requiring steroids or immune modulating medications
9. History of testing HIV positive
10. Current smoker or tobacco user
11. Current or recent history (past 6 months) of drug or alcohol abuse or dependence
12. Participation in any weight control or investigational drug study within 6 weeks of screening
13. Serious or unstable medical or psychological conditions that, in the opinion of the investigator, would compromise the subject's safety for successful study participation
14. Gastrointestinal Disorders (gallbladder disease, Crohn's disease, etc)
15. Previous weight loss surgery
16. History of bulimia or anorexia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2012-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in maternal weight from early pregnancy (< 20 weeks gestation) to 6 months and 1 year postpartum | Approximately 18 months

SECONDARY OUTCOMES:
Change in maternal weight from early pregnancy to delivery | Approximately 6 months
Change in maternal cardiometabolic biomarkers and additional anthropometrics (insulin sensitivity and secretion, fasting lipids, blood pressure, waist circumference) from early pregnancy to 6 months and 1 year postpartum | Approximately 18 months
Change in infant weight and length from birth to 6 months and 1 year of age | Approximately 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Sharon J. Herring, MD, MPH, Principal Investigator — Temple University
Locations (1):
- Temple University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Herring SJ, Cruice JF, Bennett GG, Rose MZ, Davey A, Foster GD. Preventing excessive gestational weight gain among African American women: A randomized clinical trial. Obesity (Silver Spring). 2016 Jan;24(1):30-6. doi: 10.1002/oby.21240. Epub 2015 Nov 23. PMID 26592857
- [Result] Herring SJ, Cruice JF, Bennett GG, Darden N, Wallen JJ, Rose MZ, Davey A, Foster GD. Intervening during and after pregnancy to prevent weight retention among African American women. Prev Med Rep. 2017 Jun 1;7:119-123. doi: 10.1016/j.pmedr.2017.05.015. eCollection 2017 Sep. PMID 28660118